CLINICAL TRIAL: NCT05777434
Title: Effects of Scapulothoracic Stabilization Exercises on Pain and Neck Function in Patients With Chronic Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2023/6
Record Dates: First submitted 2023-03-09; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Neck Pain
Keywords: Chronic pain, proprioception, range of motion
MeSH Terms: conditions — Neck Pain; Chronic Pain

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial having two groups. One group will receive conventional physical therapy along with cervical stabilization exercises and the second will receive Scapulothoracic Stabilization Exercises in addition to Cervical Stabilization Exercises with conventional physical therapy. Both groups will be recruited concurrently.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Conventional Physical Therapy) (Active Comparator): Patients in this group will recieve conventional physical therapy including hot pack and TENS for pain relief, axial elongtion exercises to correct posture, cervical isometrics and cervical stabilization exercises (cervical bracing with deep neck flexor activation followed by extremity ROM) along with general flexibility exercises.
  Each exercise would be performed with a hold time of 5-10 sec and 8-12 reps. A total of 12 sessions would be conducted over a period of 4 weeks.
  Interventions: Procedure: Conventional Physical Therapy for Chronic Neck Pain
- Group B (Scapulothoracic Stabilization Exercises) (Experimental): Patients will recieve scapulothoracic stabilization exercises in addition to the convential physical therapy including hot pack, TENS, axial elongation, cervical isometrics and cervical stabilization exercises. SSE would include scapular adduction and shoulder external rotation, B/L shoulder extension with scapular retraction, Eccentric scapular retraction, Brügger exercise and Forward punch. Exercises would be given using latex Thera-Band, or acc. to patient strength for mild to moderate resistance.
  Each exercise would be performed with a hold time of 5-10 sec and 8-12 reps. A total of 12 sessions would be conducted over a period of 4 weeks.
  Interventions: Procedure: Conventional Physical Therapy for Chronic Neck Pain; Procedure: Scapulothoracic Stabilization Exercises

INTERVENTIONS:
Procedure: Conventional Physical Therapy for Chronic Neck Pain — Conventional physical therapy for Chronic Neck Pain will include hot pack and TENS for pain relief, axial elongtion exercises to correct posture, cervical isometrics and cervical stabilization exercises. After 2 weeks, functional training will be added. Sets and repetitions will be increased progressively.
Procedure: Scapulothoracic Stabilization Exercises — • Scapulothoracic stabilization exercises in addition to conventional physical therapy will include scapular adduction and shoulder external rotation, B/L shoulder extension with scapular retraction, Eccentric scapular retraction, Brügger exercise and Forward punch. Exercises would be given using latex Thera-Band, or acc. to patient strength for mild to moderate resistance. After 2 weeks, functional training will be added. Sets aand repetitions will be increased progressively.
  Arms: Group B (Scapulothoracic Stabilization Exercises)

SUMMARY:
Neck pain is a common musculoskeletal disorder, involving discomfort and pain around the neck region, which results in limited neck function. Due to chronic neck pain, patient's neck function, cervical proprioception, ROM and cervical muscle strength is affected. Exercise is considered as one of the evidence-based modality to decrease pain, prevent further injury, increase muscle strength, endurance and flexibility, improve proprioception, and contribute and sustain normal life activities. In addition, recent studies suggest that exercises including not only neck but also scapulothoracic region might be more beneficial for the management of patients with chronic neck pain.Scapulothoracic stabilization exercises in addition to cervical stabilization exercises have the potential of improving this cervical sensorimotor control, however evidence is deficient Hence, this study was designed to evaluate the effectiveness of adding scapula-thoracic stabilization training to conventional physical therapy on pain and neck function in the patients with chronic neck pain.

DETAILED DESCRIPTION:
The prevalence of neck pain has increased among general population due to several factors like wroking conditions, postural abnormalitites, sedentary lifestyle, previous trauma to neck region, and altered neuromuscular control of cervical muscles, which are the main risk factors as stated in the literature. Neck pain is the second most prevalent musculoskeletal disorder and ranked 21st on global burden of disease. According to literature, it causes 30% level of restriction in performance of daily life tasks. Sleeping, driving, recreational activities and absence from work are the daily life tasks in which they face difficulty.Due to work absenties and loss of productivity can lead to reduction of quality of life of individual as well as social and ecnomical loss.

Over time, several treatment approaches have been developed to treat neck pain but the most important thing is the correction of faulty biomechanics. One such technique is scapulothoracic stabilization exercise for patients of neck pain. There are findings that support the scapular stabilization exercises for reducing neck pain and disability level.Literature reviewed regarding assessment and treatment of chronic neck pain patients revolve around pain, neck function and range of motion, however limited evidance is available on cervical proprioception and deep cervical flexors strength This research presents comparison between conventional (including TENS,hot pack and cervial focused exercises) and scapulothoracic stabilization exercises in addition to conventional treatment for chronic neck pain. It will expand current understanding of importance of scapulothoracic stabilization exercises for chronic neck pain patients in improving pain,neck function,range of motion, cervical proprioception and deep cervical flexors strength.

The main objective of this study is to compare the conventional treatment and scapulothoracic stabilization exercises along with conventional treatment in chronic neck pain patients.

The participants meeting the eligibility criteria will be recruited, followed by random allocation to 2 groups,Group A (conventional) and Group B (scapulothoracic stabilization exercises plus conventional), respectively.Both groups will recieve standard treatment protocol which conjsist of hot pack, TENS, stretchings,post isometric relaxation and home exercise plan.Twelve treatment sessions will be performed on altervative days. Pretreatment and post treatment measurements of pain, neck function, neck range of motion, cervical proprioception and deep cervical flexors strength will be noted for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Chronic neck pain greather than 3 months
* Adults aged 18-45 years
* Both Male and Female
* Subjects with non-specific neck pain without specific identifiable etiology (infection, inflammatory disease etc)

Exclusion Criteria:

* Patients with history of previous neck/ shoulder surgery
* History of cervical spine injury or surgery
* History of any psychological disorder.
* Pregnant females.
* Patient suffering from neck pain secondary to other conditions (neoplasm,neurological or vascular disease)
* Patient experiencing neck pain due to other causes such as tumors, fractures, radiculopathy etc.
* Patients who have received physiotherapy for neck pain from last 1 month

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-15 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 4 weeks
  Pain will be measured using the Visual Analog Scale (VAS)
Neck Function | 4 Weeks
  Neck function of patients will be assessed using Neck Disability Index. A higher score indicates more disability
Cervical Proprioception | 4 Weeks
  : Cervical Proprioception of patients will be assessed using Cervical Joint Position Error Test. Reposition accuracy error will be determined in Lateral flexion and rotation (right & left). A higher repositioning error indicates poor joint position sense or proprioception.
Cervical Range of Motion | 4 Weeks
  Cervical Proprioception of patients will be measured using inclinometer. Flexion, extension and lateral flexion will be measured.
Deep Cervical Flexor Strength | 4 Weeks
  Deep Cervical flexor strength of patients will be measured using CranioCervical Flexion Test in crook-lying position.

CONTACTS AND LOCATIONS:
Overall Officials: Manahil Shahid, Principal Investigator — FUI
Locations (1):
- Foundation University Islamabad, Islamabad, Federal, Pakistan